CLINICAL TRIAL: NCT00207532
Title: Dosage Effects of Folic Acid on Blood Folates of Honduran Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Ministry of Health, Honduras (Other Government); Project Healthy Children (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-4501
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Spina Bifida and Anencephaly
MeSH Terms: conditions — Neural tube defects X-linked | interventions — Folic Acid

INTERVENTIONS:
Drug: folic acid

SUMMARY:
CDC staff at the National Center on Birth Defects and Developmental Disabilities have been working closely with a Honduras-based organization, Project Healthy Children (PNS) and the Ministry of Health, on a folic acid supplementation study among female maquila workers. Participants are divided into two groups. One group receives a 1.0 milligram pill daily while the other group receives a 5.0 milligram pill weekly. The aim of this study is to assess serum blood folate levels measured at baseline, midpoint, and endpoint of the study. Hypothesis: Folic acid (5mg)given once weekly is as effective as folic acid (1mg)given daily in raising blood folate levels.

ELIGIBILITY:
Inclusion Criteria:

minimum employment in factory 6 mths

-

Exclusion Criteria:

* pregnant
* currently consuming folic acid
* prior birth-defect affected pregnancy
* chronic disease
* currently taking folic acid antagonist

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2005-03; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Milla, Principal Investigator — Project Healthy Children (Honduras)
Locations (1):
- PROTEXSA, San Pedro Sula, Honduras